CLINICAL TRIAL: NCT05496374
Title: A Randomized, Investigator-Blinded, Placebo-Controlled, Multicenter, Phase 2, Dose-Ranging Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of SPR720 as Compared With Placebo for the Treatment of Patients With Mycobacterium Avium Complex (MAC) Pulmonary Disease
Brief Title: A Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of SPR720 as Compared With Placebo for the Treatment of Participants With Mycobacterium Avium Complex (MAC) Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR720-202
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Nontuberculous Mycobacterial Pulmonary Disease (NTM-PD)
Keywords: Mycobacterium avium Complex; MAC; Pulmonary disease
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Investigator Blind: Placebo (Placebo Comparator): Participants received SPR720 matching-placebo capsules, orally, once daily (QD) for 56 days.
  Interventions: Drug: Placebo
- Investigator Blind: SPR720 500 mg (Experimental): Participants received SPR720 500 mg (250 mg × 2) capsules along with 2 SPR720 matching- placebo capsules, orally, QD for 56 days.
  Interventions: Drug: SPR720 500 mg
- Investigator Blind: SPR720 1000 mg (Experimental): Participants received SPR720 1000 mg (250 mg × 4) capsules, orally, QD for 56 days.
  Interventions: Drug: SPR720 1000 mg
- Open-label: SPR720 1000 mg (Experimental): Participants received SPR720 1000 mg (250 mg × 4) capsules, orally, QD for 56 days.
  Interventions: Drug: SPR720 1000 mg
- Open-label: SPR720 500 mg (Experimental): Participants received SPR720 500 mg (250 mg × 2) capsules, orally, twice daily (BID) for 56 days.
  Interventions: Drug: SPR720 500 mg

INTERVENTIONS:
Drug: Placebo — Placebo-matching capsules was administered orally.
  Arms: Investigator Blind: Placebo
Drug: SPR720 500 mg — SPR720 500 mg (250 mg × 2 capsules) was administered orally.
  Arms: Investigator Blind: SPR720 500 mg; Open-label: SPR720 500 mg
Drug: SPR720 1000 mg — SPR720 500 mg (250 mg × 4 capsules) was administered orally.
  Arms: Investigator Blind: SPR720 1000 mg; Open-label: SPR720 1000 mg

SUMMARY:
The purpose of the study is to evaluate

1. The microbiological response and clinical efficacy of SPR720 compared with placebo in participants with nontuberculous mycobacteria pulmonary disease (NTM-PD).
2. The safety and tolerability of SPR720 in participants with NTM- PD
3. The pharmacokinetic (PK) of SPR719, active moiety, following orally (po) administered prodrug SPR720 in participants with NTM-PD.

ELIGIBILITY:
Inclusion Criteria:

1. Has a prior diagnosis of NTM-PD due to MAC according to American Thoracic Society (ATS) criteria
2. Has at least one prior lower respiratory culture (sputum or bronchoalveolar lavage [BAL]) positive for MAC in the 12 months prior to consent
3. Has an induced sputum culture at Screening positive for MAC by quantitative culture on solid agar
4. Is either treatment naïve and has not received any prior treatment for MAC, OR if previously treated for MAC and meets all of the following criteria:

   1. Has a history of successful treatment with sputum culture conversion to negative
   2. Has recent sputum or BAL culture evidence of recurrent or relapsed disease and
   3. Has been off therapy for at least 3 months prior to consent
5. Has clinical signs and symptoms within the 6 weeks prior to consent that are consistent with NTM-PD with ≥2 of the following:

   1. chronic cough
   2. fatigue
   3. frequent throat clearing
   4. shortness of breath (dyspnea)
   5. coughing up of blood (hemoptysis)
   6. excessive mucus (sputum) production
   7. fever (temperature >38ºC or >100.4ºF)
   8. night sweats
   9. loss of appetite
   10. unintended weight loss
   11. wheezing
   12. chest pain
6. Has a measured forced expiratory volume in the first second following maximal inhalation (FEV1) % predicted ≥30% within 3 months prior to consent. If prior FEV1% predicted test result is not available, obtain FEV1% predicted at Screening to confirm eligibility

Exclusion Criteria:

1. In the opinion of the Investigator, is not a candidate for a 5-month delay in initiation of standard multidrug therapy to participate in a placebo-controlled clinical trial (e.g., participant has severe symptoms or, extensive disease burden)
2. Has disseminated or extrapulmonary NTM disease
3. Has end-stage NTM-PD or treatment-refractory NTM-PD
4. Has isolation on lower respiratory (sputum or BAL) cultures of any Mycobacterium species other than those included in MAC within the 6 months prior to consent
5. Has any other condition or prior therapy, which, in the opinion of the Investigator, would make the participant unsuitable for this study, including compliance with all study assessments and adherence to the protocol schedule of assessment
6. Prior exposure to SPR720. Participants who are unable to comply with the requirements of the study or who in the opinion of the Investigator should not participate in the study are not eligible

   * Other inclusion and exclusion criteria as per protocol may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Slope of the Weekly Sputum Log10 Colony Forming Units Per Millilitre (CFU/mL) Change From Day 1 Through 56 in micro-Intent to Treat (m-ITT) Population | Days 1 through 56 (end of the treatment [EOT])

SECONDARY OUTCOMES:
Slope of the Weekly Sputum Log10 CFU/mL Change From Days 1 Through 28 in micro-ITT Population | Days 1 through 28
Slope of the Time to Positivity (TTP) using Mycobacteria Growth Indicator Tube (MGIT) on Samples of Induced Sputum From Days 1 Through 56 (EOT) in micro-ITT Population | Days 1 through 56 (EOT)
Change from Baseline in the Sputum Log10 CFU/mL in the micro-ITT Population | Days 1 through 56 (EOT)
Change from Baseline in the Sputum TTP Using MGIT in micro-ITT Population | Days 1 through 56 (EOT)
Time to Negative Sputum Culture in micro-ITT Population | Days 1 through 56 (EOT)
Percent with Negative Sputum Culture in micro-ITT Population | Days 14 through Day 84 (FU)
Changes in Susceptibility in SPR719 From Days 1 through 56 (EOT) in the micro-ITT Population | Days 1 through 56 (EOT)
  Susceptibility is ≥4-fold increase in minimum inhibitory concentration for same pathogen identified at Baseline.
Clinical Response in the micro-ITT Population | Baseline up to Day 84 (FU)
  Investigator indicated their assessment of participants overall clinical response as resolved, improved, unchanged, or worsened.
Clinical Response in the Clinically Evaluable (CE) Populations | Baseline up to Day 84 (FU)
  Investigator indicated their assessment of participants overall clinical response as resolved, improved, unchanged, or worsened.
Change From Baseline in 11-point Nontuberculous Mycobacteria Pulmonary Disease (NTM-PD) Symptoms and Impact Scale for Quality of Life (QOL) Assessments | Baseline up to FU Day 84
  The 11-point NTM-PD Symptoms and Impact Scale will evaluate specific clinical signs and symptoms and QOL improvements and will include symptoms of chronic cough, fatigue, frequent throat clearing, dyspnea, hemoptysis, excessive mucus (sputum) production, chills, night sweats, loss of appetite, unintended weight loss, wheezing, and chest pain.
Change From Baseline in 6-point Patient Global Impression of Severity (PGI-S) Scale for Quality of Life (QOL) Assessments | Baseline up to FU Day 84
  The PGI-S scale is comprised of a 6-point verbal descriptor scale to determine meaningful change reported for the other symptom ratings in participants with NTM-PD.
Change From Baseline in 7-point Patient Global Impression of Change (PGI-C) scale for Quality of Life (QOL) Assessments | Baseline up to FU Day 84
  The PGI-C scale is a patient-reported rating of improvement on a 7-point verbal descriptor scale.
Change From Baseline in Flu, COVID-19, or Other Illness Questionnaire (2 questions) for Quality of Life (QOL) Assessments | Baseline up to FU Day 84
  This 2-question form will assess the participants flu, COVID-19 or other illness status and how these illnesses have affected the participants NTM-PD disease over the past 7 days.
Change from Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS®) V1.0 Fatigue Short form 7a scale for Quality of Life (QOL) Assessments | Baseline up to FU Day 84
  The PROMIS® scale will assess the participants experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities using a validated 5-point Likert scale.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | From first dose of study drug (Day 1) up to follow up Day 84
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational/experimental) product, whether related to this product or not.
Maximum Plasma Concentration (Cmax) (Intensive PK group only) | Pre-dose and post-dose on Days 1 and 14
Time to reach Cmax (Tmax) (Intensive PK group only) | Pre-dose and post-dose on Days 1 and 14
Area Under the Concentration-time Curve (AUC0-τ) (Intensive PK group only) | Pre-dose and post-dose on Days 1 and 14
Accumulation Ratio of SPR719 Cmax on Day 14 Compared to Day 1 (Intensive PK group only) | Pre-dose and post-dose on Days 1 and 14
Accumulation Ratio of SPR719 AUC0-τ on Day 14 Compared to Day 1 (Intensive PK group only) | Pre-dose and post-dose on Days 1 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Xilla Ussrey, MD, Study Director — Spero Therapeutics Inc
Locations (28):
- United States (28):
  - Medical Facility, Birmingham, Alabama
  - Medical Facility, Fresno, California
  - Medical Facility, Los Angeles, California
  - Medical Facility, Newport Beach, California
  - Medical Facility, Northridge, California
  - Medical Facility, Santa Clarita, California
  - Medical Facility, Washington D.C., District of Columbia
  - Medical Facility, Kissimmee, Florida
  - Medical Facility, Loxahatchee Groves, Florida
  - Medical Facility, Miami, Florida
  - Medical Facility, Sebring, Florida
  - Medical Facility, Tampa, Florida
  - Medical facility, Atlanta, Georgia
  - Medical Facility, Iowa City, Iowa
  - Medical Facility, Kansas City, Kansas
  - Medical Facility, New Bedford, Massachusetts
  - Medical Facility, Rochester, Minnesota
  - Medical Facility, Lebanon, New Hampshire
  - Medical Facility, New Hyde Park, New York
  - Medical Facility, Chapel Hill, North Carolina
  - Medical Facility, Winston-Salem, North Carolina
  - Medical Facility, Cleveland, Ohio
  - Medical Facility, Portland, Oregon
  - Medical Facility, Pittsburgh, Pennsylvania
  - Medical Facility, Charleston, South Carolina
  - Medical Facility, Denison, Texas
  - Medical Facility, Sherman, Texas
  - Medical Facility, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No